CLINICAL TRIAL: NCT03878225
Title: The Ketone Mono Ester Study - Does a Ketogenic Dietary Supplement Reduce Alcohol Withdrawal Symptoms in Humans
Brief Title: Does a Ketogenic Dietary Supplement Reduce Alcohol Withdrawal Symptoms in Humans?
Acronym: KME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Dmsc,, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-18045204
Record Dates: First submitted 2019-02-13; First posted 2019-03-18 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal; Ketosis
MeSH Terms: conditions — Alcoholism; Ketosis

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, placebo controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be stratified according to gender and body-weight. The randomization uses stratified permuted block randomization. Selected un-blinded personnel will carry out the randomization procedure. After randomization is carried out, the ketone mono ester or placebo beverages will be delivered to the patients by blinded personnel. Patients, investigators, other caregivers and persons performing data analysis will remain blinded from the time of randomization until the time of database unlock. Un-blinded project personnel will prepare and pack the ketone mono ester/placebo beverage in identical bottles. The placebo beverage will consist of water added with a colorless, bitter flavor enhancer (Bitrex®) and a sweetening agent (Stevia) to approximate the taste of the ketone mono ester beverage as closely as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Mono Ester (Active Comparator): The ketone mono ester is commercially available dietary supplement beverage named "H.V.M.N. Ketone Ester", marketed by HVMN Inc®. The KME beverage consists of water, D-β-hydroxybutyrate ester, stevia leaf extract, natural flavors, malic acid, potassium sorbate and potassium benzoate. The active ingredient is the D-β-hydroxybutyrate ester, with each dose containing 25g. Participants will be asked to ingest this 5 times daily for 3 days (72 hours), to a total of 15 doses during the study.
  Interventions: Dietary Supplement: H.V.M.N. Ketone Ester
- Placebo (Placebo Comparator): The placebo beverage will consist of water added with a colorless, bitter flavor enhancer and a sweetening agent (Stevia) to approximate the taste of the KME beverage as closely as possible. The bitter flavor enhancer used is denatonium benzoate (Bitrex®). The placebo beverage will be delivered to patients in bottles identical to those used in the active arm. Patients, investigators and other caregivers will be blinded to treatment allocation until time of database unlock.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: H.V.M.N. Ketone Ester — The ketone mono ester will be ingested 5 times daily for 3 days (72 hours). Please see above for details.
  Other Names: Ketone beverage, ketone mono ester (https://hvmn.com/ketone)
  Arms: Ketone Mono Ester
Other: Placebo — The placebo will be ingested 5 times daily for 3 days (72 hours). Please see above for details.
  Arms: Placebo

SUMMARY:
A ketogenic diet (KD) is high in fat and low in carbohydrates and induces ketosis. KD is an approved non-pharmacological therapy for drug-resistant child epilepsy. Research has shown that a KD can reduce the behavioral measures of alcohol withdrawal symptomatology in rats. Ketosis is also possible to achieve without adherence to a KD, by ingestion of a ketogenic dietary supplement. In this study, we want to investigate if the attenuating effect of the KD observed in rodents, is also applicable in humans, i.e. whether a ketogenic dietary supplement, here a ketone monoester, would be effective in suppressing alcohol withdrawal symptoms in humans.

Objective:

To test the effect of a ketogenic dietary supplement on the need for benzodiazepines in managing alcohol withdrawal syndrome in humans.

Eligibility:

Adults 18-70 years who are alcohol dependent and are seeking treatment for alcohol withdrawal syndrome in an out-patient setting.

Design:

Double blinded, randomized clinical trial. The participants will be randomized to receive either the ketone ester beverage, or a placebo beverage.

The study will be conducted over three days (72 hours), with follow-up at 1 month and 1 year after completion. A sub-set of patients will undergo Magnetic Resonance Spectroscopy (MRS) following withdrawal treatment, and again after 1 month.

DETAILED DESCRIPTION:
Neuroimaging studies have shown that acute alcohol administration decreases glucose metabolism in the human brain, which was initially thought to reflect decreased brain function. However, subsequent studies showed that even low doses of alcohol, with minimal behavioral effects, also decreased baseline brain glucose metabolism and further. This led to the hypothesis that the reduction in brain glucose metabolism during alcohol intoxication reflected the brain's utilization of an alternate energy substrate, e.g. the alcohol metabolite acetate. Acetate is not a ketone body, but biochemically similar to the ketone bodies, which include acetoacetate, BHB and acetone. Ketone bodies are similarly taken up by the Monocarboxylate Transporters in neurons, and other brain tissue. A pre-clinical trial has demonstrated that the implementation of a KD for 10 days significantly reduced the behavioral measures of alcohol withdrawal symptomatology in rats. In this study, we want to investigate if the attenuating effect of the KD observed in rodents, is also applicable in humans, i.e. whether a ketogenic dietary supplement, here a ketone monoester, would be effective in suppressing alcohol withdrawal symptoms in humans.

Objectives:

We will investigate the effect of a five times daily oral administration of a ketone dietary supplement beverage vs. placebo on the need for benzodiazepines in alcohol withdrawal syndrome. The KME beverage is a supplement to standardized out-patient alcohol withdrawal treatment.

Study population:

36 participants aged 18-70 with a diagnosis of alcohol use disorder according to the DSM-V, ICD-10, and a previous history of treatment-requiring alcohol withdrawal syndrome.

Design:

Clinical double-blinded, randomized, placebo-controlled, three-day clinical trial, with an MRS (Magnetic Resonance Spectroscopy) sub-study. The participants will be randomized to receive either the ketone ester beverage, or a placebo beverage 5 times daily. Participants will be asked to register benzodiazepine use in a medication-diary during the study. Participants will be asked to self-monitor blood-glucose and ketone levels by use of fingerstick measurements. During the study patients will be evaluated for withdrawal severity, and complete questionnaires on alcohol craving, sleep, anxiety and mood.

ELIGIBILITY:
Inclusion Criteria KME trial

1. Between 18 and 70 years of age.
2. Ability to provide written informed consent as determined by the physical examination and verbal communication. The capacity to consent will be determined by study personnel.
3. Alcohol-dependent individuals must meet alcohol dependency syndrome criteria according to ICD-10 and alcohol use disorder according to DSM-5, have a score >15 on the Alcohol Use Disorder Identification Test (AUDIT) and a history of previous treatment for alcohol withdrawal syndrome following cessation of alcohol use.

Inclusion Criteria Healthy Volunteers for MRS sub-study

1. Between 18 and 70 years of age.
2. Ability to provide written informed consent as determined by the physical examination and verbal communication. The capacity to consent will be determined by study personnel.
3. Light drinkers (LD): Alcohol consumption less than 7 drinks per week typically over the past year and no more than three drinks per occasion. AUDIT score below 7 in the Alcohol Use Disorder Identification Test.
4. Heavy drinkers (HD): Not treatment-seeking and not fulfilling criteria for alcohol dependence syndrome according to ICD-10 or alcohol use disorder according to DSM-5. For at least one-year consuming alcohol at a typical rate of above a level of 14 drinks per week for men and consume at least 4 drinks per day at least once per week. For females, consume alcohol in excess of 11 drinks per week and exceed 3 drinks per day at least once per week.
5. Long term sober (LTS): For the long-term sober group, a previous diagnosis of alcohol dependence, consumed no alcohol in the previous 6 months.

Exclusion Criteria KME trial and MRS sub-study

1. Diagnosis of current psychiatric disorder that is deemed not stable by the study physician, except for the following:

   * Diagnosis of nicotine dependence
   * Alcohol withdrawal patients may have a diagnosis of alcohol dependence
   * HD may have a diagnosis of alcohol abuse
2. Lifetime diagnosis of bipolar disorder, schizophrenia, paranoid psychosis or mental retardation.
3. Incapable of understanding and/or speaking Danish.
4. Head trauma with loss of consciousness for more than 60 minutes (self-report, medical history).
5. Lifetime diagnosis of epilepsy.
6. Alcohol withdrawal seizures within the previous 3 months.
7. Use of any medication that could interfere with study assessments, including anticonvulsants, benzodiazepines and non-benzodiazepine hypnotics (Zopiclone and/or Zolpidem). Use of medications will be reviewed by a study physician on a case by case basis.
8. Body Mass Index, BMI, < 18.5 kg/m2 or body weight <60 kg or >120kg.
9. Urine positive for cocaine, amphetamines, methadone, opioids or benzodiazepines.
10. Blood glucose >12.2 mmol/L on finger-prick measurement (>7.0 if over-night fasted).
11. Known kidney disease, pancreatic disease, porphyria or other mitochondrial diseases, type 1 diabetes, type 2 diabetes or any other history of severe somatic illness that the investigator believes would interfere with trial participation.
12. Known cirrhosis or clinical evidence of significant liver disease, such as ascites or hepatosplenomegaly.
13. Following a low-carbohydrate diet, intermittent fasting diet or consuming nutritional ketone supplements.
14. Other substance use dependency than alcohol and/or nicotine and/or cannabis within the previous 1 month.
15. Benzodiazepine dependence within the previous 1 month and/or use of benzodiazepines within the previous 14 days.
16. Females of childbearing potential who are pregnant, breast-feeding or have intention of becoming pregnant within the next 4 months, or are not using contraceptives (during the whole study period) considered as highly effective (combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) intrauterine device - IUD, IUS, bilateral tubal occlusion, vasectomized partner, sexual abstinence) (HMA - Clinical Trials Facilitation and Coordination Group, 2014).
17. Participated in a clinical trial with investigational medication or weight reduction within the previous three months.
18. Use of Disulfiram (Antabus) in the previous 14 days prior to any planned KME ingestion or MRS procedure.
19. For HD and LD groups in MRS sub-study only: Inability to abstain from alcohol for 24 hours, to reduce risks and to avoid confounding results with alcohol withdrawal.
20. For HD and LD in MRS sub-study only: History of alcohol use disorder or alcohol withdrawal symptoms requiring medication
21. For participants undergoing MRS (all HD, LD, and LTS, some KME patients): Implanted metallic devices or objects that could potentially prove harmful when exposed to the MRS environment or procedures. Patients in the alcohol withdrawal group can still participate in the KME study if meeting this criterion, but cannot undergo subsequent MRS.
22. Any condition that the investigator estimates would interfere with trial participation and/or the safety of the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Benzodiazepine use | 2 years
  Quantity of benzodiazepine needed to manage alcohol withdrawal symptoms.
Magnetic Resonance Spectroscopy sub-study | 2 years
  For the MRS sub-study brain BHB, GABA and Glutamate will be measured with 1H MRS following KME ingestion. Results will be compared with healthy volunteers with differing alcohol consumption habits.

SECONDARY OUTCOMES:
Sleep quality | 2 years
  Daily self-reported sleep quality on a VAS scale. Self-reported estimated sleep-time in previous 24 hours.
Alcohol withdrawal symptoms. | 2 years
  Alcohol withdrawal symptoms assessed by use of the revised Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar). Measures of pulse, blood pressure and respiratory frequency.
Anxiety | 2 years
  Anxiety assessed with VAS questionnaires
Alcohol craving | 2 years
  Alcohol craving assessed with the Desire for Alcohol Questionnaire (DAQ)
Alcohol intake | 2 years
  Asses alcohol intake after the trial at one month and one year after completion, using the Timeline Follow Back method (TLFB). Assess the Alcohol Use Disorder Identification Test (AUDIT) at the beginning of the trial and one year after termination of the trial
Mood | Assess mood measured by VAS questionnaires during the trial, and by the Major Depressive Inventory (MDI) at screening and one-month follow-up
  Mood, assessed by the Major Depression Inventory scale, MDI. The MDI is a self report mood questionnaire. Symptoms are rated based on how the patient has been feeling over the past two weeks.
  The diagnostic demarcation line indicates at which point a symptom is severe enough to be used in the DSM-IV diagnostic algorithm of major depression.
  Each question has a point giving system from 0-5 points. The higher the score, the more severe outcome. Scores from 20-24 indicates minor depressive symptoms. Scores from 25-29 indicates a moderate depression. Scores from 30 and above indicates major depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, MD, DMSc, Principal Investigator — Psychiatric Center Copenhagen, Rigshospitalet
Locations (2):
- Denmark (2):
  - Novavi Lyngby, Lyngby, Danmark (DK)
  - Psychiatric Center Copenhagen, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bornebusch AB, Mason GF, Tonetto S, Damsgaard J, Gjedde A, Fink-Jensen A, Thomsen M. Effects of ketogenic diet and ketone monoester supplement on acute alcohol withdrawal symptoms in male mice. Psychopharmacology (Berl). 2021 Mar;238(3):833-844. doi: 10.1007/s00213-020-05735-1. Epub 2021 Jan 7. PMID 33410985